CLINICAL TRIAL: NCT03386448
Title: The Safety and Efficacy of Naltrexone and Scopolamine Utilized in Combination in the Treatment of Major Depression: A Double Blinded, Randomized, Controlled Pilot Study
Brief Title: The Safety and Efficacy of Naltrexone and Scopolamine Utilized in the Treatment of Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Taub Group (Industry)
Responsible Party: Principal Investigator, Neal Taub MD, Principle Investigator, The Taub Group
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 701
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Scopolamine; Naltrexone

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized, controlled parallel design
Who Masked: Participant, Care Provider
Masking Description: The participants and physician are both blinded to medication vs. control medication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): Participants will receive placebo medication
  Interventions: Drug: placebo arm
- Active (Experimental): participants will receive active medications scopolamine and naltrexone
  Interventions: Drug: Scopolamine and naltrexone

INTERVENTIONS:
Drug: Scopolamine and naltrexone — participants will receive scopolamine and naltrexone in buccal drops
  Arms: Active
Drug: placebo arm — participants will receive placebo medications
  Arms: control

SUMMARY:
The purpose of this clinical trial is to determine the safety and efficacy of scopolamine utilized in conjunction with naltrexone for the treatment of major depression.

DETAILED DESCRIPTION:
The study will be a double blinded, randomized controlled trial. The medications will be administered orally. The sample size will be 40 participants, 20 in the treatment group and 20 in the control group. The study period will be 4 weeks. Eligible participants will have major depression by history for at least 8 weeks, between 18-65 years old, and in generally good health other than depression. The MADRS questionaire will be utilized to determine the response to the medications.

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged 18-65
* in good health other than major depression for 8 weeks or more
* negative pregnancy test
* able to comply with instructions
* able to provide informed consent

Exclusion Criteria:

* pregnant or lactating
* danger to self or others
* severe kidney or liver disease
* schizophrenia
* allergy to scopolamine or naltrexone
* glaucoma
* Monoamine oxidase (MAO) inhibitor use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Taub, Principal Investigator — The Taub Group
Locations (1):
- The Taub Group, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control(Placebo): Participants will receive placebo medication
  placebo arm: participants will receive placebo medications
- Active(Scopolamine and Naltrexone): participants will receive active medications scopolamine and naltrexone. Scopolamine dose was 0.15mg BID and naltrexone dose was 1mg BID for 4 weeks.
  Scopolamine and naltrexone: participants will receive scopolamine and naltrexone in buccal drops
Period: Overall Study
Arm/Group | Control(Placebo) | Active(Scopolamine and Naltrexone)
Started | 6 | 8
Completed | 6 | 6
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control(Placebo) | Active(Scopolamine and Naltrexone) | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 8 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Response to Medications as Assessed by Change in Score on Modified MDRS Scale From Baseline to End of Study Period
Description: The Montgomery-Asberg (MADRS) depression scale will be utilized throughout the study. The scale is scored 0-60, 0 signifying no depression symptoms and 60 signifying very severe depression. A diagnosis of depression will be given to a participant in this study for a MADRS score of 20 or greater. A clinical response to medication will be noted when a participant has a 25% or greater decrease in MADRS score during the trial.
Time Frame: Baseline and 4 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Control(Placebo) | Active(Scopolamine and Naltrexone)
Number analyzed (Participants) | 6 | 6
units on a scale | 3.5 [1 to 7] | 12.5 [6 to 23]
Statistical Analysis 1: Comparison: Control(Placebo) vs Active(Scopolamine and Naltrexone); Test type: Superiority — Student test was performed; p = 0.03, t-test, 2 sided; Mean Difference (Final Values) = 9.0

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events for 8 weeks.
Arm/Group | Control(Placebo) | Active(Scopolamine and Naltrexone)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control(Placebo) (N=6) | Active(Scopolamine and Naltrexone) (N=8)
Nausea (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT03386448/Prot_SAP_000.pdf